CLINICAL TRIAL: NCT07363876
Title: The Efficacy of Ultrasonication in Combination With Corticosteroid Intraarticular Injection for Arthritis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Principal Investigator, Kuo-Lung Lai, Principal Investigator, Taichung Veterans General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TCVGH-1150801B; CF25511A (Other: TCVGH IRB)
Record Dates: First submitted 2026-01-08; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-12

CONDITIONS: Arthritis; Ultrasonication; Intra-articular Injections; Rheumatology
MeSH Terms: conditions — Arthritis | interventions — Ultrasonic Therapy; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ultrasonication in combination with corticosteroid intraarticular injection (Experimental)
  Interventions: Device: Therapeutic Ultrasound; Procedure: Intra-articular corticosteroid injection
- corticosteroid intraarticular injection (Active Comparator)
  Interventions: Procedure: Intra-articular corticosteroid injection

INTERVENTIONS:
Device: Therapeutic Ultrasound — Therapeutic Ultrasound (TUS) is a non-invasive treatment widely used in physical medicine and rehabilitation for musculoskeletal conditions. Since its introduction in the mid-20th century, TUS has gained popularity in clinical practice due to its ability to penetrate tissues, target treatment areas precisely, and exhibit minimal side effects. This study aims to investigate the mechanisms of action, clinical efficacy, and safety of therapeutic ultrasound in musculoskeletal therapy.
  Arms: ultrasonication in combination with corticosteroid intraarticular injection
Procedure: Intra-articular corticosteroid injection — Injection of triamcinolone (3-50 mg depending on joint size) into the affected joint. Administered once per participant.

SUMMARY:
This study investigates whether ultrasound therapy applied prior to intra-articular corticosteroid injection can enhance the treatment efficacy for patients with joint arthritis and assess its safety. Adult patients diagnosed with arthritis in the limbs who are indicated for corticosteroid injection are eligible, while patients with joint replacement, hip joint involvement, gout, infectious arthritis, or local cellulitis are excluded.

Ultrasound therapy is a valuable physical therapy tool for musculoskeletal diseases, producing therapeutic effects through thermal and non-thermal mechanisms. It can improve tissue extensibility, reduce joint stiffness, increase local blood flow, enhance metabolism during tissue repair, and facilitate drug absorption. This study evaluates whether applying ultrasound before intra-articular corticosteroid injection improves therapeutic outcomes in patients with arthritis, and assesses the safety of this combined intervention. Patients aged 18 or older, diagnosed with limb arthritis, and indicated for corticosteroid injection are eligible. Exclusion criteria include joint replacement, hip joint involvement, gout, infectious arthritis, or local cellulitis at the treatment site.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older.
* Diagnosed with arthritis in the limbs.
* Inadequate response to or contraindication for oral anti-inflammatory medications.
* Assessed by a physician as requiring intra-articular corticosteroid injection.

Exclusion Criteria:

* History of joint replacement (prosthetic joint) in the affected area.
* Hip joint involvement.
* Diagnosis of gout.
* Infectious arthritis.
* Presence of cellulitis at the treatment site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12-29 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Reduction in Synovial Swelling Area Assessed by Joint Ultrasound | From enrollment to the end of treatment at 2 weeks
  Synovial swelling area (pixels) assessed by joint ultrasound. A treatment response is defined as a ≥50% reduction in synovial swelling area from baseline.
Change in Power Doppler (PD) Score of the Target Joint | From enrollment to the end of treatment at 2 weeks
  Power Doppler (PD) score (range 0-3) of the target joint assessed by joint ultrasound. A treatment response is defined as a PD score of 0 at 2 weeks post-treatment.
Change in Pain Visual Analogue Scale (VAS) | From enrollment to the end of treatment at 2 weeks
  Pain intensity assessed using a visual analogue scale (VAS 0-10). A treatment response is defined as a ≥50% reduction in VAS score from baseline or a VAS score ≤1 at 2 weeks post-treatment.

SECONDARY OUTCOMES:
Absence of Synovitis Recurrence Based on Power Doppler (PD) Score | From enrollment to 3 months post-treatment
  Absence of synovitis recurrence assessed by Power Doppler (PD) ultrasound. Recurrence is defined as any increase in PD score compared with the 2-week post-treatment assessment.
Absence of Synovial Swelling Recurrence on Gray-Scale Ultrasound | From enrollment to 3 months post-treatment
  Absence of synovial swelling recurrence assessed by gray-scale ultrasound. Recurrence is defined as an increase in synovial swelling area of ≥20% compared with the 2-week post-treatment assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Kuo-Lung Lai, MD, Principal Investigator — Taichung Veterans General Hospital (TaichungVGH)